CLINICAL TRIAL: NCT01948401
Title: A STUDY TO MEASURE SERUM PERIOSTIN, ASTHMA-RELATED BIOMARKERS AND RESPONSE TO PREDNISOLONE IN ADULT AND ADOLESCENT PATIENTS WITH SEVERE ORAL CORTICOSTEROID-DEPENDENT ASTHMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: WB28850
Record Dates: First submitted 2013-09-06; First posted 2013-09-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Adrenal Cortex Hormones; Prednisolone

ARMS (3):
- Controlled asthma (Experimental)
  Interventions: Drug: LABA; Drug: corticosteroids
- Uncontrolled asthma with additional OCS (Experimental)
  Interventions: Drug: LABA; Drug: corticosteroids; Drug: prednisolone
- Uncontrolled asthma without additional OCS (Experimental)
  Interventions: Drug: LABA; Drug: corticosteroids

INTERVENTIONS:
Drug: LABA — long-acting beta-agonist treatment
Drug: corticosteroids — chronic treatment with oral corticosteroids, high dose inhaled corticosteroids
Drug: prednisolone — additional 0.5 mg/kg orally for 7 days
  Arms: Uncontrolled asthma with additional OCS

SUMMARY:
This interventional, open study will evaluate clinical data in relation to biomarkers in patients 12 to 75 years of age with severe oral corticosteroid (OCS) - dependent asthma. Patients with uncontrolled asthma will be offered an additional escalation of OCS at a dose of 0.5 mg/kg for 7 days. Patients enrolled in this study would be eligible to be enrolled in a future placebo-controlled intervention study designed to measure the steroid-sparing effect of lebrikizumab.

ELIGIBILITY:
Inclusion Criteria:

* Adult and adolescent patients , >/=12 to </=75 years of age at the time of informed consent
* Severe asthma (as defined by GINA step 5 classification of asthma severity) after a detailed systematic assessment (the BTS UK Difficult Asthma Network assessment model [Heaney et al 2010] or equivalent) and follow-up by an asthma specialist for at least six months
* History of asthma treatment with high doses of inhaled corticosteroids (ICS ) (>/=1500 mcg beclomethasone dipropionate daily, or equivalent) and long-acting beta-2 agonists (LABAs), with or without an additional controller, for at least six months before Screening
* Chronic treatment with maintenance oral corticosteroids (OCS) for at least six months before the time of informed consent ; (baseline OCS dose: adults 10 to 40 mg/day, adolescents 5 to 40 mg/day daily dose equivalent)
* Compliance with OCS therapy will be based on prior detectable levels of serum prednisolone, cortisol suppression, or observation of Cushingoid appearance consistent with regular systemic steroid use
* Diagnosis of refractory asthma (Heaney et al 2010) with OCS dependence on minimal effective or maximum tolerated dose
* Confirmed (by chest x-ray) absence of other significant lung disease
* Documented history of bronchodilator reversibility response of >/=12% and >/=200 mL within the past 12 months before the time of informed consent

Exclusion Criteria:

* Baseline FEV1 </=39% of predicted
* Asthma exacerbation (as defined by protocol) within 28 days before the time of informed consent or during Screening
* Major episode of infection requiring admission to hospital for >/=24 hours or treatment with intravenous antibiotics within the 28 days before the time of informed consent or during Screening or requiring treatment with oral antibiotics within the 14 days before the time of informed consent or during Screening
* Active parasitic infection or Listeria monocytogenes infection within the 6 months before the time of informed consent
* For adults active tuberculosis (TB) requiring treatment within the 12 months before the time of informed consent (patients are also required to have no recurrence of symptoms in the 12 months following completion of TB treatment), or for adolescents history of active TB requiring treatment
* Known history of severe clinically significant immunodeficiency
* Evidence of acute or chronic hepatitis or known liver cirrhosis
* Inadequate liver function
* Diagnosis or history of malignancy, or current investigation for possible malignancy
* Other clinically significant medical disease that is uncontrolled despite treatment or that is likely, in the opinion of the investigator, to require a change in therapy or affect the ability to participate in the study
* Current smoker or former smoker with a smoking history of >15 pack-years
* Current use of an immunomodulatory/immunosuppressive therapy or past use within three months or five drug half-lives (whichever is longer) before the time of informed consent
* Use of a biologic therapy (including omalizumab) at any time during the 4 months before the time of informed consent
* History of anaphylaxis with omalizumab treatment or history of anaphylaxis to any therapeutic biological agent
* Use of zileuton or roflumilast at any time during the two months before the time of informed consent
* Initiation of or change in allergen immunotherapy within three months before the time of informed consent
* Treatment with an investigational agent within 30 days of informed consent or 5 half-lives of the investigational agent, whichever is longer
* Pregnant or lactating women
* Body mass index (BMI) >38 kg/m2
* Body weight <40 kg

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Serum periostin levels | up to 95 days

SECONDARY OUTCOMES:
Asthma quality of life questionnaire for adults and adolescents aged 12 years and older (AQLQ12+) | up to 95 days
IL-13 related biomarker levels | up to 95 days
Lung function: Forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) | up to 95 days
Safety: Incidence of adverse events | up to 95 days
Patient reported outcomes: Asthma Control Questionnaire (ACQ-7) | up to 95 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United Kingdom (9):
  - Belfast
  - Birmingham
  - Glasgow
  - Hampshire
  - Leicester
  - London
  - Manchester
  - Newcastle upon Tyne
  - Nottingham

REFERENCES:
- [Derived] Busby J, Holweg CTJ, Chai A, Bradding P, Cai F, Chaudhuri R, Mansur AH, Lordan JL, Matthews JG, Menzies-Gow A, Niven R, Staton T, Heaney LG. Change in type-2 biomarkers and related cytokines with prednisolone in uncontrolled severe oral corticosteroid dependent asthmatics: an interventional open-label study. Thorax. 2019 Aug;74(8):806-809. doi: 10.1136/thoraxjnl-2018-212709. Epub 2019 Apr 2. PMID 30940770